CLINICAL TRIAL: NCT03395054
Title: The Effects of Cervical Stabilization Exercises on Pulmonary Functions and Respiratory Muscle Strength in Patients With Neck Pain
Brief Title: The Effects of Cervical Stabilization Exercises on Pulmonary Functions and Respiratory Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, birgül morkoç, principal investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 151623-09
Record Dates: First submitted 2017-11-22; First posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Neck Pain
Keywords: neck pain; pulmonary function test; respiratory muscle strength; cervical stabilization exercises
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the stabilization group (Other): the stabilization group performed cervical stabilization exercises in lying, sitting, standing and on a swisball 3times a week during 8 weeks.
  Interventions: Other: cervical stabilization exercises
- the control group (Other): the control group performed conventional exercises including neck isometric, isotonic and posture exercises 3 times a week during 8 weeks.
  Interventions: Other: conventional exercises

INTERVENTIONS:
Other: cervical stabilization exercises — cervical stabilization exercises
  Arms: the stabilization group
Other: conventional exercises — conventional exercises
  Arms: the control group

SUMMARY:
This study aims to assess the effects of stabilization exercises on pulmonary functions and respiratory muscle strength. 42 participants with neck pain enrolled the study.

DETAILED DESCRIPTION:
This study aims to assess the effects of stabilization exercises on pulmonary functions and respiratory muscle strength. 42 participants with neck pain enrolled the study. Participants were divided into two groups, stabilization group (n=21) and the control group (n=21). The participants underwent a total of 24 sessions of treatment thrice a week for eight weeks under the supervision of a physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* neck pain longer than 3 months
* patients between ages of 18 and 55

Exclusion Criteria:

* patients with neurologic symptoms
* patients with chronic pulmonary disease
* previous surgery on cervical region

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
pulmonary functions | 8 weeks
  pulmonary functions were measured with spirometric tests by two experienced physical therapists.
respiratory muscle strength | 8 weeks
  respiratory muscle strength was measured using mouth pressure device by two experienced physical therapists.

CONTACTS AND LOCATIONS:
Overall Officials: Birgül Morkoç, phd student, Principal Investigator — Hacettepe University
Locations (1):
- Institute of Health Sciences, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
none are planned to be shared